CLINICAL TRIAL: NCT00694499
Title: Retrospective Single Centre Study Which Investigates the Safety of the Non-Operative Management of Patients With High Grade Blunt Liver Injuries (NOMLI) and the Impact of to the LI Collateral Intra- and Extra-Abdominal Damage on Interventions and Outcome
Brief Title: Non-Operative Management of High Grade Blunt Hepatic Injury: Clinical Complications and the Role of Collateral Damage
Acronym: NOMLI
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Beat Schnüriger,MD, Dep. of Visceral and Transplant Surgery, Bern University Hospital
Other Study IDs: KEK 29_04_2008
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Liver Injury
Keywords: Morbidity; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients with blunt liver injury

SUMMARY:
Little is known about the role of collateral damage in patients with high grade liver injuries (LI). This retrospective single centre study investigates the safety of the non-operative management of patients with high grade blunt liver injuries (NOMLI) and the impact of to the LI collateral intra- and extra-abdominal damage on interventions and outcome. We first hypothesized that NOMLI can be safely achieved also in high-grade liver injured patients, the management of trauma patients with LI mainly consist of the treatment of collateral damages and their complications, and causes of death are in the majority of cases not liver related. A retrospective study involving 183 patients with blunt hepatic injuries was therefore carried out to investigate these hypotheses.

DETAILED DESCRIPTION:
Background:

Modern approach to liver injured patients favours non-operative management of liver injury (NOMLI) including endovascular artery occlusion. Numerous studies over the past two decades have confirmed the feasibility of NOMLI in up to 95% of hemodynamically stable patients with blunt trauma mechanisms. To further improve the outcome of patients with hepatic injuries, investigations should focus on the overall morbidity and mortality of NOMLI. Purely hepatic-related complication rates in most series are low, ranging from 0-7% and parallel the grade of liver lesion. But the majority of patients included in those studies suffered low-grade liver injuries (LI). Regarding the safety of NOMLI in high grade lesions, the results may be biased. Complications in patients with high-grade LI are more frequent and their management is considerably more complex. Regarding the sparsely available literature focussing on the morbidity of NOMLI in high grade LI, hepatic-related complication rates of 11 and 13% have been described. Only the LI grade and the amount of packed red blood cell (PRBC) transfusion at 24 hours postinjury predicted hepatic-related complications. No data is available concerning the impact of collateral intra- and extra-abdominal damage on complications of NOMLI in those patients. Of note, up to 75% of patients with LI suffer from collateral intra- and extra-abdominal lesions. These injuries vary in their surgical importance but severe complications and to the LI independent laparotomies must be expected in a significant number of patients. Rates of such nonspecific laparotomies have been described in up to 20% of patients with hepatic trauma. Over the past decade, overall mortality of liver injured patients remained relatively constant, averaging between 10-15%. This mortality rate represents deaths of all causes in the clinical course of these complex trauma patients. There are studies which already suggested, that early deaths in patients with LI also were caused by uncontrolled bleedings from associated intra- and extra-abdominal injuries, and that most late deaths result from collateral head injuries and sepsis with multi-organ-failure (MOF). But no detailed data about the occurrence of extra-abdominal complications after NOMLI has been published so far.

Objective:

We first hypothesized that NOMLI can be safely achieved also in high-grade liver injured patients, the management of trauma patients with LI mainly consist of the treatment of collateral damages and their complications, and causes of death are in the majority of cases not liver related. A retrospective study involving 183 patients with blunt hepatic injuries was therefore carried out to investigate these hypotheses.

Methods:

The study was conducted at the Bern University Hospital, Switzerland between January 2000 and December 2006. An average of 286 (range, 204-344) multiple injured patients were treated in our level I trauma centre each year. Only blunt liver injured patients were included. All charts (including surgery and autopsy reports) were reviewed retrospectively. Demographic data collected included age, gender, mechanism of injury. Injury patterns were defined by the Abbreviated Injury Score (AIS) and Injury Severity Score (ISS). The grade of hepatic injury was determined by an experienced radiologist and by two experienced hepatobiliary surgeons in parallel based on contrast enhanced computed tomography (CT) scan findings (Siemens® Somatom Sensation 16) or by laparotomy according to the American Association for the Surgery of Trauma Organ Injury Scale for hepatic injuries. For the current study, high-grade injuries were considered grades 3 to 5. Other data collected included the number and types of surgical procedures, hepatic-related and overall complications, and causes of deaths. All patients were managed and resuscitated using the protocols outlined in the Advanced Trauma Life Support (ATLS) manual of the American College of Surgeons Committee on Trauma. NOMLI was

ELIGIBILITY:
Inclusion Criteria:

* Patients with blunt liver injury
* Treated from 2000-2006 at Bern University Hospital

Exclusion Criteria:

* < 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with blunt liver injury treated at Bern University Hospital from 2000-2006
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2000-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Morbidity | During primary in-hospital stay

SECONDARY OUTCOMES:
Liver-related morbidity | During in-hospital stay
Other morbidity | During in-hospital stay
Mortality | During in-hospital stay
Surgical interventions needed | During in-hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Inderbitzin, MD, Study Director — Dep. of Visceral and Transplant Surgery, Bern University Hospital Bern
Locations (1):
- Dep. of Visceral and Transplant Surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] John TG, Greig JD, Johnstone AJ, Garden OJ. Liver trauma: a 10-year experience. Br J Surg. 1992 Dec;79(12):1352-6. doi: 10.1002/bjs.1800791238. PMID 1486439
- [Background] Velmahos GC, Toutouzas K, Radin R, Chan L, Rhee P, Tillou A, Demetriades D. High success with nonoperative management of blunt hepatic trauma: the liver is a sturdy organ. Arch Surg. 2003 May;138(5):475-80; discussion 480-1. doi: 10.1001/archsurg.138.5.475. PMID 12742948
- [Background] Pachter HL, Knudson MM, Esrig B, Ross S, Hoyt D, Cogbill T, Sherman H, Scalea T, Harrison P, Shackford S, et al. Status of nonoperative management of blunt hepatic injuries in 1995: a multicenter experience with 404 patients. J Trauma. 1996 Jan;40(1):31-8. doi: 10.1097/00005373-199601000-00007. PMID 8576995
- [Background] Kozar RA, Moore FA, Cothren CC, Moore EE, Sena M, Bulger EM, Miller CC, Eastridge B, Acheson E, Brundage SI, Tataria M, McCarthy M, Holcomb JB. Risk factors for hepatic morbidity following nonoperative management: multicenter study. Arch Surg. 2006 May;141(5):451-8; discussion 458-9. doi: 10.1001/archsurg.141.5.451. PMID 16702516
- [Background] Kozar RA, Moore JB, Niles SE, Holcomb JB, Moore EE, Cothren CC, Hartwell E, Moore FA. Complications of nonoperative management of high-grade blunt hepatic injuries. J Trauma. 2005 Nov;59(5):1066-71. doi: 10.1097/01.ta.0000188937.75879.ab. PMID 16385280
- [Background] Gao JM, Du DY, Zhao XJ, Liu GL, Yang J, Zhao SH, Lin X. Liver trauma: experience in 348 cases. World J Surg. 2003 Jun;27(6):703-8. doi: 10.1007/s00268-003-6573-z. Epub 2003 May 13. PMID 12733001
- [Background] Hurtuk M, Reed RL 2nd, Esposito TJ, Davis KA, Luchette FA. Trauma surgeons practice what they preach: The NTDB story on solid organ injury management. J Trauma. 2006 Aug;61(2):243-54; discussion 254-5. doi: 10.1097/01.ta.0000231353.06095.8d. PMID 16917435
- [Background] Resources for optimal care of the injured patient: an update. Task Force of the Committee on Trauma, American College of Surgeons. Bull Am Coll Surg. 1990 Sep;75(9):20-9. No abstract available. PMID 10106239
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394
- [Background] Cogbill TH, Moore EE, Jurkovich GJ, Feliciano DV, Morris JA, Mucha P. Severe hepatic trauma: a multi-center experience with 1,335 liver injuries. J Trauma. 1988 Oct;28(10):1433-8. PMID 3172301